CLINICAL TRIAL: NCT04837989
Title: Diabetes Body Project: Effectiveness of a Virtually Delivered Eating Disorder Prevention Program Among Young Females With Type 1 Diabetes
Brief Title: Effectiveness of the Diabetes Body Project Among Females With Type 1 Diabetes
Acronym: DBP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Data will be written up as a pilot RCT study and experiences and results will inform the start of a multi-site trial
Sponsor: Oslo University Hospital (Other)
Collaborators: The Dam Foundation (Other); Norwegian Diabetes Association (Other)
Responsible Party: Principal Investigator, Line Wisting, Researcher, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6860
Record Dates: First submitted 2021-03-29; First posted 2021-04-08 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Feeding and Eating Disorders; Diabetes Mellitus, Type 1; Body Image
MeSH Terms: conditions — Feeding and Eating Disorders; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes Body Project (Experimental): Participants randomized to the experimental condition will receive virtual Diabetes Body Project groups immediately.
  Interventions: Behavioral: Diabetes Body Project
- Educational (Active Comparator): Participants randomized to the control condition will receive an education brochure and will be offered the Diabetes Body Project after 6 months.
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Diabetes Body Project — Six virtually delivered Diabetes Body Project groups over six weeks (one hour a week); 5-6 participants and 2 group facilitators
  Arms: Diabetes Body Project
Behavioral: Psychoeducation — Individuals assigned to the psychoeducational control condition will receive an educational brochure, and complete similar assessments and assessment time points as the experimental condition. Individuals in the control group will be offered Diabetes Body Project group participation after six months.
  Arms: Educational

SUMMARY:
Young females with type 1 diabetes (T1D) is at high risk of eating disorders (ED), with prevalence rates of ED more than double those of non-diabetes peers. T1D and ED are both associated with serious somatic complications, and when occurring together the prognosis is even worse. Despite the frequency and severity of this comorbidity, there is a lack of intervention studies and no consensus on how to best prevent and treat this comorbidity. To remedy this, we have developed a virtual diabetes-adapted version of the ED prevention program Body Project, i.e. the Diabetes Body Project. This study examines the effectiveness of the Diabetes Body Project to reduce ED risk factors and symptoms among young females with T1D.

DETAILED DESCRIPTION:
Type 1 Diabetes (T1D) T1D is caused by an autoimmune destruction of the insulin-producing beta cells in the pancreas, leading to complete lack of insulin. Insulin is necessary to regulate blood glucose levels. T1D is a national and international health challenge and priority, and Norway has among the highest incidence of T1D in the world. This is a growing problem (incidence in Norway has increased by 30% in the last 15 years) with profound long-term complications due to sub optimal metabolic control, including atherosclerosis, with subsequent cerebrovascular and cardiovascular disease, retinopathy, neuropathy and nephropathy.

Significant rates of psychological problems are associated with T1D. One study investigated young patients with T1D and found that 11% screened positive for depression, 21% for anxiety, and 21% for disordered eating. Patients with a positive screen had twice the odds of having poor metabolic control (high HbA1c) as those without. Other psychological correlates reported to influence T1D self-care and metabolic control include illness perceptions, attitudes to insulin, and quality of life.

Eating disorders and Disturbed Eating Behaviors (DEB) ED affect approximately 5% of the female Norwegian population between the ages of 15-44 years, and onset is most common during adolescence. ED are characterized by disordered eating such as restricted intake or bingeing and purging, a morbid preoccupation with food, weight and shape and major disturbances in cognition with distortion of body image. The main eating disorders as defined in the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) are Anorexia Nervosa (AN), Bulimia Nervosa (BN), Binge Eating Disorder (BED), and Otherwise Specified Feeding and Eating Disorders (OSFED). A large amount of disturbed eating behaviors do not meet full criteria for the diagnoses described above and is often referred to as sub-clinical eating problems or disturbed eating behaviors. The term "disturbed eating behavior" (DEB) is used here to refer to sub-clinical eating problems.

Comorbid T1D and DEB Numerous studies indicate that T1D is a risk factor for the development of DEB. Possible mediating factors include weight loss accompanying disease onset, weight gain with the initiation of insulin treatment, dietary restraint as part of diabetes management, and the deliberate insulin under dosing or omission as an effective weight loss strategy. However, few longitudinal studies of comorbid T1D and DEB exist, and there is a lack of knowledge about the specific risk factors for the development of DEB in T1D. One recent longitudinal study states that DEB was common and persistent in their sample of adolescent females with T1D. At the 14-year follow-up, a total of 32% met criteria for a current eating disorder, and DEB was reported in 59% of the participant, confirming the severity of this comorbidity. The cumulative probability of onset was 60% by the age of 25 years.

DEB is common and persistent in young women with T1D, with prevalence rates double those of non-diabetic populations. Our prior study found that the prevalence of DEB was 27% among young Norwegian girls with T1D, indicating that these comorbidities are common in Norway. Comorbid T1D and DEB are associated with poor metabolic control and increased rates of morbidity and mortality. For example in Nielsen's study of comorbid T1D and anorexia nervosa, the mortality rate at 10 years follow-up was 2.5 % for T1D and 6.5% for anorexia nervosa; though when comorbid it rose to 35%. DEB also poses a risk of serious physical complications, thereby contributing to much poorer prognosis.

The nature of T1D-specific DEB It has been suggested that the nature of DEB in T1D is specific and qualitatively different from DEB in non-diabetes populations. It is hypothesized that a diabetes-specific DEB has its origins in the nature and course of T1D and T1D treatment. T1D constitutes a considerable burden on the young patients and their families. The continuous self-regulation task of adjusting insulin dose to diet, physical activity and emotional state to maintain blood glucose levels according to recommendations is accompanied by the threat of developing serious diabetes late complications. Such factors may contribute to increased weight- and shape concerns among patients with T1D (particularly females). Reducing or omitting insulin is an efficient weight loss strategy uniquely available to individuals with diabetes, but is associated with increased morbidity and mortality. In addition to insulin restriction, bulimic features such as binge eating and self-induced vomiting or misuse of laxatives are common symptoms of DEB in T1D.

Despite the frequency and severity of comorbid T1D and DEB/ED, there is a lack of studies on how to prevent this condition. The Body Project is reported to be the most effective ED prevention program in the general population, but this has not been tested in a T1D population. The overall aim of this study is therefore to evaluate a diabetes-adapted version of the ED prevention program the Body Project (i.e. the Diabetes Body Project) among young females with T1D. Specifically, we hypothesize that the Diabetes Body Project can improve i) ED risk factors (i.e. thin beauty ideal internalization, body dissatisfaction, and dietary restraint) and symptoms (ED measure composite score); ii) blood glucose control (i.e. Hemoglobin A1c and time in range); and iii) diabetes-specific psychological aspects (i.e. diabetes distress and illness perceptions) relative to an educational condition.

ELIGIBILITY:
Inclusion Criteria:

* Female, 16-35 years, type 1 diabetes, acknowledges at least some level of body image concerns

Exclusion Criteria:

* Other forms of diabetes, males

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
The Ideal-Body Stereotype Scale-Revised (IBSS-R) | Baseline, change from baseline to 6 weeks, change from baseline to 6-months
  Thin beauty ideal internalization, scores range from 1-5, higher scores indicate higher levels of internalization
The Body Parts Scale | Baseline, change from baseline to 6 weeks, change from baseline to 6-months
  Nine items on body dissatisfaction, scores range from 1-5, higher scores indicate more body dissatisfaction
Dietary restraint | Baseline, change from baseline to 6 weeks, change from baseline to 6-months
  Eating restriction, scores range from 1-5, higher scores indicate more eating restriction
The Diabetes Eating Problem Survey - Revised | Baseline, change from baseline to 6 weeks, change from baseline to 6-months
  Total score to indicate level of eating disorder psychopathology, scored 0-5, higher scores indicate higher levels of eating disorder psychopathology
Social attitudes towards appearance questionnaire (SATAQ) 4R | Baseline, change from baseline to 6 weeks, change from baseline to 6-months
  Appearance pressures and internalization, answers range from 1-5, higher scores indicate more pressures/internalization
Social Comparison Scale | Baseline, change from baseline to 6 weeks, change from baseline to 6-months
  The degree to which individuals compare themselves to others, score 1-10, higher scores indicate more favorable social compariso

SECONDARY OUTCOMES:
Blood glucose control | Baseline, change from baseline to 6 weeks, change from baseline to 6-months
  Hemoglobin A1c (HbA1c) and time in range. Higher HbA1c indicate poorer blood glucose control. Higher time in range indicate better blood glucose control
Problem Areas in Diabetes (PAID) | Baseline, change from baseline to 6 weeks, change from baseline to 6-months
  Diabetes distress, scored 0-4, higher scores indicate higher degree of diabetes distress
Brief Illness Perception Questionnaire | Baseline, change from baseline to 6 weeks, change from baseline to 6-months
  Diabetes illness perceptions, scores range from 0-10, higher scores indicate more threatening/negative of their diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Line Wisting, PhD, Principal Investigator — Oslo University Hospital, Division of Mental Health and Addiction
Locations (1):
- Oslo Unviersity Hospital, Oslo, Norway